CLINICAL TRIAL: NCT04891926
Title: Influence of Hormonale Changes on Diuresis and LUTS in the Gynaecological Population
Brief Title: Hormonal Influences on Diuresis
Acronym: HODI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EC2014/1241
Record Dates: First submitted 2021-05-04; First posted 2021-05-19 (Actual); Last update posted 2021-05-19 (Actual); Status verified 2021-04

CONDITIONS: Nocturia; Menopause; LUTS; Diuresis
MeSH Terms: conditions — Nocturia | interventions — Hematologic Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hormonal therapy (Experimental): Patients choosing to start hormoanl treatment using ural or transdermal estrogen.
  Interventions: Diagnostic Test: ICIQ FLUTS Questionaires; Diagnostic Test: Frequency Volume Chart; Diagnostic Test: Renal Function Profile; Diagnostic Test: Blood Analysis

INTERVENTIONS:
Diagnostic Test: ICIQ FLUTS Questionaires — Questionnaire observing the impact on voiding disfunctions
Diagnostic Test: Frequency Volume Chart — Frequency Volume Chart measures the voided volumes and fluid intake during 3 days in order to observe patients bladder capacity, total and nighttime voided volume and voiding frequency
Diagnostic Test: Renal Function Profile — The RFP is a 24-hour urine analysis in which urine samples are collected at fixed time points every 3 hours, starting 3 hours after the first morning void. This RFP was collected on a separated day to the FVC. Daytime samples were taken between 10:00-11:30 (U1), 13:00-15:30 (U2), 16:00-17:30 (U3), 19:00-20:30 (U4), and 22:00-23:30 (U5). The night-time samples were taken between 1:00-2:30 (U6), 4:00-5:30 (U7) and 7:00-8:30 (U8), and the volume of each interim void, was noted to calculate the 24h, daytime and night-time urine volume and diuresis rate. On each of this 8 samples, creatinine, osmolality, sodium and urea concentration were analysed. Subsequently, the renal clearance of creatinine, solutes, sodium and potassium (Usubst x Uflow / Psubst) and FWC (urine flow - solute clearance) were calculated.
Diagnostic Test: Blood Analysis — Blood analysis in order to observ postmenopausal state, osmolalitity and sodium.

SUMMARY:
The aim of this study was to observe the effect of hormonal treatment (oral or transdermal substitution therapy) on diuresis (salt and water diuresis) and lower urinary tract symptoms (LUTS) in postmenopausal women

ELIGIBILITY:
Inclusion Criteria:

* Patients in a postmenopausal state wo wanted to start treatment for menopausal symptoms (hot flushes etc)

Exclusion Criteria:

-

Min Age: 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Menopausal women
Enrollment: 70 (Actual)
Dates: Start 2015-05-01; Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Change of HT on nocturnal frequency | 6 months
  Change of nocturnal frequency by 1 nocturnal void after 6 months of hormonal treatment.

SECONDARY OUTCOMES:
Effect on nocturnal urine production | 6 months
  Change of the nocturnal urine production by hormonal treatment by the volume of one micturition (+- 200ml)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Pauwaert K, Bruneel E, Van Laecke E, Depypere H, Everaert K, Goessaert AS. Does hormonal therapy affect the bladder or the kidney in postmenopausal women with and without nocturnal polyuria: Results of a pilot trial? Maturitas. 2022 Jun;160:61-67. doi: 10.1016/j.maturitas.2022.01.009. Epub 2022 Jan 29. PMID 35550708